CLINICAL TRIAL: NCT05367115
Title: National Cheng Kung University Hospital
Brief Title: Verification of the Epidemiology and Mortality of Rare Diseases in Taiwan With Real-world Evidence
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Chih-Hsing Wu, Associate Professor, National Cheng-Kung University Hospital
Other Study IDs: Taiwan rare diseases
Record Dates: First submitted 2022-05-02; First posted 2022-05-10 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Rare Diseases; Epidemiology; Morbidity; Morality; Comorbidities and Coexisting Conditions; Health Care Utilization
MeSH Terms: conditions — Rare Diseases; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Familial Amyloidotic Polyneuropathy: The Familial Amyloidotic Polyneuropathy patients are validated in the catastrophic illness certification.
  Interventions: Other: longitudinal observational study
- Osteogenesis imperfecta: The Osteogenesis imperfecta patients are validated in the catastrophic illness certification.
  Interventions: Other: longitudinal observational study
- (Acute Hepatic) Porphyria: The (Acute Hepatic) Porphyria patients are validated in the catastrophic illness certification.
  Interventions: Other: longitudinal observational study

INTERVENTIONS:
Other: longitudinal observational study — longitudinal observational study

SUMMARY:
This study aims to explore the longitudinal incidence and prevalence trends of selected muscular and bone-related rare diseases, i.e., Familial Amyloidotic Polyneuropathy (FAP), Primary hyperoxaluria, Wilson's disease, Cystic fibrosis, Osteogenesis imperfecta, Porphyria, and Primary Paget disease, and analyze healthcare utilization.

DETAILED DESCRIPTION:
A rare disease (RD) means any disease that affects a small percentage of the population. According to the "Rare Disease and Orphan Drug Act" in 2000, RD is defined as the prevalence of lower than 10,000 people in Taiwan, or with special circumstances, and announced after review by the "Review Committee for Rare Diseases and Orphan Drugs". There are many different causes of RD, such as genetic and infection. Although researchers have made progress in learning how to diagnose, treat, and even prevent a variety of RD, but there is still much to do because most rare diseases have no treatments. Due to the low morbidity rate and fewer numbers of people who suffer from RD, patients have been impacted by a severe pathology and insufficiently recognized, diagnosed, and cured. However, prevalence, healthcare utilization, and economic impacts of rare diseases based on real-world evidence are still unknown in the world, especially in Taiwan. In 2020, there were 226 diseases officially proclaimed as RD and 17,592 patients in Taiwan, and approved 108 orphan drugs and 40 special nutrients for treating those patients to reduce their financial burden.

ELIGIBILITY:
Inclusion Criteria:

* The RD patients were defined as at least two ambulatory care records or one inpatient record in one year with Familial Amyloidotic Polyneuropathy (FAP), Osteogenesis imperfecta, and Acute Hepatic Porphyria between 2009 and 2017.

Exclusion Criteria:

* The RD patients were diagnosed with Familial Amyloidotic Polyneuropathy (FAP), Osteogenesis imperfecta, and Acute Hepatic Porphyria before 2009.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The rare disease patients are validated in the Taiwan catastrophic illness certification.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Number of incidences | 12 years
  The number of new cases had diagnosed with Familial Amyloidotic Polyneuropathy (FAP), Primary hyperoxaluria, Wilson's disease, Cystic fibrosis, Osteogenesis imperfecta, Porphyria, and Primary Paget disease during the time of observation from Taiwan's National Health Insurance Research Database.
Number of prevalence | 12 years
  The number of participants who have had diagnosed with Familial Amyloidotic Polyneuropathy (FAP), Primary hyperoxaluria, Wilson's disease, Cystic fibrosis, Osteogenesis imperfecta, Porphyria, and Primary Paget disease during the time of observation from Taiwan's National Health Insurance Research Database.
Number of death | 12 years
  The number of participants who have had diagnosed with Familial Amyloidotic Polyneuropathy (FAP), Primary hyperoxaluria, Wilson's disease, Cystic fibrosis, Osteogenesis imperfecta, Porphyria, and Primary Paget disease with death during the time of observation from Taiwan's National Death Registry.
Number of Health Care Utilization | 12 years
  The health care use from Taiwan's National Health Insurance Research Database in participants who have had diagnosed with Familial Amyloidotic Polyneuropathy (FAP), Primary hyperoxaluria, Wilson's disease, Cystic fibrosis, Osteogenesis imperfecta, Porphyria, Primary Paget disease during the time of observation.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hsing Wu, MD, Study Director — National Cheng Kung University
Locations (1):
- Department of Family Medicine, National Cheng Kung Univ Hosp, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No